CLINICAL TRIAL: NCT01996371
Title: Radiographic and Clinical Outcomes Following Unilateral or Bilateral Posterior Fixation in Minimally Invasive Transforaminal Lumbar Interbody Fusions
Brief Title: Radiographic and Clinical Outcomes Following Unilateral or Bilateral Posterior Fixation in MI-TLIF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: H Francis Farhadi, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, H Francis Farhadi, MD, PhD, Assistant Professor, Ohio State University
Organization: Ohio State University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2013H0171
Record Dates: First submitted 2013-11-01; First posted 2013-11-27 (Estimated); Results first posted 2021-11-09 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-10

CONDITIONS: Lumbar Disease
MeSH Terms: conditions — Disease | interventions — Pedicle Screws

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 (Other): Unilateral pedicle screws
  Interventions: Device: Pedicle Screw
- Group 2 (Other): Ipsilateral pedicle screws, contralateral facet screw
  Interventions: Device: Pedicle Screw
- Group 3 (Other): Bilateral pedicle screws
  Interventions: Device: Pedicle Screw

INTERVENTIONS:
Device: Pedicle Screw

SUMMARY:
The purpose of this study is to compare the healing of the patients spine at 24-months following surgery and screw placement among 3 groups. The doctor will also compare clinical outcomes and the immediate and delayed medical and surgical complications among the 3 study groups. The goal of this study is to determine if treating patients with one of the 3 groups is better than the others.

DETAILED DESCRIPTION:
Patient must be between 18 and 80 years old and have problems with the bones in there lower back (lumbar disease) for which Cautious management over at least 3 months has not brought relief from back and/or leg pain. Patients will be scheduled to undergo surgery to treat there lumbar disease. The surgery will be followed by placement of screws in the back of the bones of there lower back. This includes placing solid metal rods that are connected and secured to adjacent vertebrae (bones of the back) using screws. The screws are used to hold the spine together. Everyone who takes part in this study will be assigned to one of the following 3 study groups: 1) One-sided screw placement into the bones above and below the area where the nerve is being surgically relieved of its pinching; 2) Same as group 1 but with an additional stand alone screw which crosses the spinal joint placed into the joint on the other side; 3) Screw placement on both sides into the bones above and below the area where the nerve is being surgically relieved of its pinching.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years.
* Symptomatic single-level lumbar disease including lumbosacral junction.
* Unilateral leg-dominant pain non-responsive to conservative management with concordant imaging findings. These include degenerative spondylolisthesis (grade 1 or 2), facet arthropathy +/- lateral disc herniation, recurrent disc herniation, or large central disc herniation.
* Back pain of confirmed discogenic origin (single level disease only).
* Failed conservative management for a minimum of 3 months.
* Negative serum pregnancy test (for women of childbearing potential)

Exclusion Criteria:

* Severe bilateral leg symptoms.
* Prior instrumented arthrodesis at any lumbar level.
* History of osteoporosis.
* Co-morbidities requiring medication that may interfere with bone or soft tissue healing (i.e., oral or parenteral glucocorticoids, immunosuppressive agent, methotrexate).
* Severe co-morbidities (e.g., heart, respiratory, or renal disease).
* Recent (<3 yrs) Co-incident spinal tumor or infection.
* Greater than single level symptomatic involvement.
* Associated thoracolumbar kyphotic or scoliotic deformity (>10).
* Morbid obesity (BMI > 40).
* History of metal sensitivity/foreign body sensitivity.
* Concurrent involvement in another investigational drug or device study that could confound study data.
* History of substance abuse (recreational drugs, prescription drugs, or alcohol) that could interfere with protocol assessments and/or with the subject's ability to complete the protocol required follow-up.
* Subjects who are pregnant or plan to become pregnant in the next 24 months.
* Prisoner.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-01; Primary Completion 2020-05 (Actual); Study Completion 2020-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: H. Francis Farhadi, MD, PhD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State Unviersity, Columbus, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: Unilateral: Unilateral pedicle screws
  Pedicle Screw
- Group 2: Ipsilateral: Ipsilateral pedicle screws, contralateral facet screw
  Pedicle Screw
- Group 3: Bilateral: Bilateral pedicle screws
  Pedicle Screw
Period: Overall Study
Arm/Group | Group 1: Unilateral | Group 2: Ipsilateral | Group 3: Bilateral
Started | 5 | 4 | 6
Completed | 5 | 4 | 6
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All subject ethnicity: White
Groups:
- Group 1: Unilateral pedicle screws
  Pedicle Screw
- Group 2: Ipsilateral pedicle screws, contralateral facet screw
  Pedicle Screw
- Group 3: Bilateral pedicle screws
  Pedicle Screw
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Group 3 | Total
Number analyzed (Participants) | 5 | 4 | 6 | 15
Age, Customized [Count of Participants; unit: Participants]
  Age: Age: 18-59 | 3 | 2 | 4 | 9
  Age: Age 60-80 | 2 | 2 | 2 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 3 | 5
  Male | 3 | 4 | 3 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 4 | 6 | 15
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 4 | 6 | 15

OUTCOME MEASURES:

1. Primary Outcome: Compare Bony Fusion Rates Radiographically Using CT Scans
Description: Primary Outcome: To compare bony fusion rates at two years among the three study arms, using the Brantigan, Steffee and Fraser scale. Post-operative CT scans will be evaluated at 24 months for evidence of new solid osseous trabeculations bridging across the interspace.
Time Frame: 24 months
Population: Research has been discontinued. Data not collected and therefore not analyzed.
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Bony Fusion Rates Compared Clinically Using the Visual Analog Scale (VAS) Survey
Description: To compare clinical outcomes among the three study arms utilizing the Visual Analog Scale (VAS) survey. Visual analog scales will be used to assess neck, back, arm, and leg pain. Scores can range from 0 - 10 with higher scores indicating higher levels of pain.
Time Frame: 3 months, 6 months, 12 months, 24 months
Population: Research has been discontinued. Data not collected and therefore not analyzed.
Arm/Group | Group 1: Unilateral | Group 2: Ipsilateral | Group 3: Bilateral
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Bony Fusion Rates Compared Clinically Using the Oswestry Disability Index v2 (ODI v2) Survey
Description: To compare clinical outcomes among the three study arms utilizing the Oswestry Disability Idex (ODI) survey. This survey will be used to assess how back pain affects patients' ability to function in everyday life. Scores can range from 0% to 100% with higher scores indicating higher levels of disturbance in everyday life.
Time Frame: 3 months, 6 months, 12 months, 24 months
Population: Research has been discontinued. Data not collected and therefore not analyzed.
Arm/Group | Group 1: Unilateral | Group 2: Ipsilateral | Group 3: Bilateral
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Bony Fusion Rates Compared Clinically Using the Short Form 36 Health Survey v2 (SF-36 v2)
Description: To compare clinical outcomes among the three study arms utilizing the Short Form 36 Health Survey (SF-36). This survey will be used to assess patients' physical and mental health. Scores range from 0 to 100 with higher scores indicating better physical and mental health.
Time Frame: 3 months, 6 months, 12 months, 24 months
Population: Research has been discontinued. Data not collected and therefore not analyzed.
Arm/Group | Group 1: Unilateral | Group 2: Ipsilateral | Group 3: Bilateral
Number analyzed (Participants) | 0 | 0 | 0

5. Other Pre Specified Outcome: Safety Outcome: Immediate and Delayed Medical and Surgical Complications Compared Among the Three Arms
Description: Immediate and delayed medical and surgical (including neurological) complications among the three study arms will be compared.
Time Frame: post-surgery, 6 weeks, 3 months, 6 months, 12 months, 24 months
Population: Research has been discontinued. Data not collected and therefore not analyzed.
Arm/Group | Group 1: Unilateral | Group 2: Ipsilateral | Group 3: Bilateral
Number analyzed (Participants) | 0 | 0 | 0

6. Other Pre Specified Outcome: Exploratory Outcome: Compare Bony Fusion Rates Using X-ray Based Classification Scale
Description: Comparison of bony fusion rates at 12 and 24 months among the three study arms, using an X-ray based classification scale.
Time Frame: 12 months and 24 months
Population: Research has been discontinued. Data not collected and therefore not analyzed.
Arm/Group | Group 1: Unilateral | Group 2: Ipsilateral | Group 3: Bilateral
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Enrollment to 24 Months post surgery
Arm/Group | Group 1 | Group 2 | Group 3
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/4 | 0/6
Serious Adverse Events (participants affected / at risk) | 1/5 | 1/4 | 1/6
Other Adverse Events (participants affected / at risk) | 2/5 | 2/4 | 4/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=5) | Group 2 (N=4) | Group 3 (N=6)
Compression Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) — Required surgical repair
Bilateral PEs (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) — Subject self presented to hospital with SOB-Dyspnea leading to a diagnosis of bilateral PEs. Subject transferred and admitted to ED
Disc Herniation (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) — Patient called in with increased back and leg pain after lifting a washing machine. The CNP advised imaging studies (X-rays and MRI) leading to a diagnosis of a disc herniation.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=5) | Group 2 (N=4) | Group 3 (N=6)
Acute Chronic Back and/or Leg Pain (Nervous system disorders) | 1 (1) | 1 (1) | 3 (3) — When appropriate treated with Valium and/or ESIs or no treatment
Allergic Reaction to dilaudid (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) — Intubated- Medical Management
ED Visit - Bronchitis/asthma attack (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) — Given Prednisone
RTC Impingement (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) — ESIs
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) — Narcan given

LIMITATIONS AND CAVEATS:
This study is being ended early due to low enrollment. No analysis is planned due to the small cohort.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-08-08): https://cdn.clinicaltrials.gov/large-docs/71/NCT01996371/Prot_SAP_000.pdf
  • Informed Consent Form (2017-04-11): https://cdn.clinicaltrials.gov/large-docs/71/NCT01996371/ICF_001.pdf